CLINICAL TRIAL: NCT04734054
Title: Evaluation of Pain, Discomfort, and Functional Impairments During the Orthodontic Treatment of Skeletal Maxillary Constriction Using Rapid Versus Slow Maxillary Expansion in the Early Permeant Dentition: A Randomized Controlled Trial
Brief Title: Pain, Discomfort, and Functional Impairments During Rapid and Slow Maxillary Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2021
Record Dates: First submitted 2021-01-24; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Maxillary Constriction
Keywords: posterior crossbite; rapid maxillary expansion; slow maxillary expansion; pain; discomfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid maxillary expansion (Experimental): The rapid maxillary expansion will be conducted using bonded modified Hyrax palatal expander. The expander will be activated twice daily (0.4 mm) until an overcorrection of 2-3 mm will be gained.
  Interventions: Device: Modified Hyrax Palatal Expander
- Slow maxillary expansion (Active Comparator): The slow maxillary expansion using a removable plate with a midline screw will be accomplished. The expander will be activated twice weekly until an overcorrection of 2-3 mm will be gained.
  Interventions: Device: Removable Palatal Expander

INTERVENTIONS:
Device: Modified Hyrax Palatal Expander — The rapid maxillary expansion will be performed. The expansion should be accomplished between 10 to 15 days at most. The screw is going to be turned in a rapid manner.
  Arms: Rapid maxillary expansion
Device: Removable Palatal Expander — The slow maxillary expansion will be performed. The expansion will be performed in a slow manner. Patients may need between 6 to 8 months to achieve the required expansion.
  Arms: Slow maxillary expansion

SUMMARY:
This study will assess and compare the levels of pain, discomfort, and functional impairments between rapid and slow maxillary expansion in treating skeletal maxillary constriction in the early adolescence period (i.e. between 12 and 16 years).

The study sample will consist of 32 patients who suffer from a skeletal posterior crossbite. The sample will be allocated randomly into two groups: RME group and SME group.

The patients will be asked to fill out the attached questionnaires at three assessment times.

DETAILED DESCRIPTION:
Skeletal maxillary constriction is a popular orthodontic malocclusion that can be seen at any age. The maxillary expansion is the most important treatment choice of this skeletal problem in the upper jaw. There are many types of maxillary expansion regarding the force amount and the number of expansion times: slow maxillary expansion (SME) rapid maxillary expansion (RME), and semi-rapid maxillary expansion (SRME).

Practitioners are conscious that complaints submitted by children and adolescents during the active phase of expansion, such as pain, discomfort and oral ulcers are common symptoms. This trial of two parallel groups will compare the pain, discomfort and functional impairments accompanying the rapid and slow maxillary expansion in early adolescent patients.

RME group: A bonded modified Hyrax palatal expander will be applied. SME group: A removable palatal expansion appliance with a midline screw will be applied.

To assess the pain, discomfort and functional impairments, patients will be asked to fill out questionnaires of six questions: 1) What is the degree of pain/discomfort you have experienced?; 2) Do you have difficulty in mastication?; 3) Do you have difficulty in swallowing?; 4) Do you have a sense of tension or pressure in soft tissue?; 5) Do you have swelling in soft tissue?; and 6) How easy is the treatment procedure?.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the early permanent dentition
2. Chronological age between 12 and 16 years
3. The presence of a functional unilateral posterior crossbite (with a functional shift) or bilateral posterior crossbite (without any functional shift)
4. Skeletal bilateral maxillary constriction (symmetric constriction) were assessed clinically then confirmed radiographically
5. Dental and skeletal class I and II malocclusion
6. Normal and mild vertical growth pattern
7. The presence of upper first premolars and molars
8. No general problems
9. Good oral health
10. No previous orthodontic treatment.

Exclusion Criteria:

1. Presence of periodontal diseases
2. Presence of general diseases, syndromes or cleft lip and palate
3. Patients with previous orthodontic treatment
4. Patients with severe horizontal growth pattern

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain and discomfort | T1: on the 1st day; T2: on the 7th day in the RME group and in the 3rd or 4th month in the SME group; T3: on the 15th day in the RME group and between the 6th and 8th month in the SME group
  Patients will be asked this question about their feeling of pain and discomfort (Item no 01):
  'What is the degree of pain/discomfort you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the Visual Analogue Scale (VAS) which is a 10-cm horizontal line with two focal points at its beginning and end (0: there is no pain - 10: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the difficulty in mastication | T1: on the 1st day; T2: on the 7th day in the RME group and in the 3rd or 4th month in the SME group; T3: on the 15th day in the RME group and between the 6th and 8th month in the SME group
  Patients will be asked this question about any difficulty in mastication (Item no 02):
  'Do you have difficulty in mastication?' A standardized questionnaire will assess pain, discomfort and functional impairments' levels during the active phase of treatment. The 4-point Likert scale will be used consisting of: (no), (mild), (moderate) or (severe). The patient will be asked to choose one of the four options.
Change in the difficulty in swallowing | T1: on the 1st day; T2: on the 7th day in the RME group and in the 3rd or 4th month in the SME group; T3: on the 15th day in the RME group and between the 6th and 8th month in the SME group
  Patients will be asked this question about any difficulty in swallowing (Item no 03):
  'Do you have difficulty in swallowing?' A standardized questionnaire will assess pain, discomfort and functional impairments' levels during the active phase of treatment. The 4-point Likert scale will be used consisting of: (no), (mild), (moderate) or (severe). The patient will be asked to choose one of the four options.
Change in the sensation of tension or pressure on soft tissue | T1: on the 1st day; T2: on the 7th day in the RME group and in the 3rd or 4th month in the SME group; T3: on the 15th day in the RME group and between the 6th and 8th month in the SME group
  Patients will be asked this question about any sense of tension or pressure on soft tissue (Item no 04):
  'Do you have a sense of tension or pressure in soft tissue ' A standardized questionnaire will assess pain, discomfort and functional impairments' levels during the active phase of treatment. The 4-point Likert scale will be used consisting of: (no), (mild), (moderate) or (severe). The patient will be asked to choose one of the four options.
Change in the degree of swelling in soft tissues | T1: on the 1st day; T2: on the 7th day in the RME group and in the 3rd or 4th month in the SME group; T3: on the 15th day in the RME group and between the 6th and 8th month in the SME group
  Patients will be asked this question about any swelling in soft tissue (Item no 05):
  'Do you have swelling in soft tissue?' A standardized questionnaire will assess pain, discomfort and functional impairments' levels during the active phase of treatment. The 4-point Likert scale will be used consisting of: (no), (mild), (moderate) or (severe). The patient will be asked to choose one of the four options.
Change in patient's perception of treatment ease | T1: on the 1st day; T2: on the 7th day in the RME group and in the 3rd or 4th month in the SME group; T3: on the 15th day in the RME group and between the 6th and 8th month in the SME group
  Patients will be asked this question about the ease of the treatment procedure (Item no 06):
  'How easy is the treatment procedure?' A standardized questionnaire will assess pain, discomfort and functional impairments' levels during the active phase of treatment. The 4-point Likert scale will be used consisting of: (easy), (medium), (hard) or (very hard). The patient will be asked to choose one of the four options.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rabah, DDS,MSc, Principal Investigator — Specialist and Clinical Lecturer, Department of Orthodontics, University of Damascus; Heba M Al-Ibrahim, DDS, Principal Investigator — MSc student in Orthodontics, University of Damascus, Dental School, Damascus, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus, Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martina R, Cioffi I, Farella M, Leone P, Manzo P, Matarese G, Portelli M, Nucera R, Cordasco G. Transverse changes determined by rapid and slow maxillary expansion--a low-dose CT-based randomized controlled trial. Orthod Craniofac Res. 2012 Aug;15(3):159-68. doi: 10.1111/j.1601-6343.2012.01543.x. Epub 2012 Mar 27. PMID 22812438
- [Background] Gecgelen M, Aksoy A, Kirdemir P, Doguc DK, Cesur G, Koskan O, Ozorak O. Evaluation of stress and pain during rapid maxillary expansion treatments. J Oral Rehabil. 2012 Oct;39(10):767-75. doi: 10.1111/j.1365-2842.2012.02330.x. Epub 2012 Jul 11. PMID 22783926
- [Background] Cossellu G, Lanteri V, Lione R, Ugolini A, Gaffuri F, Cozza P, Farronato M. Efficacy of ketoprofen lysine salt and paracetamol/acetaminophen to reduce pain during rapid maxillary expansion: A randomized controlled clinical trial. Int J Paediatr Dent. 2019 Jan;29(1):58-65. doi: 10.1111/ipd.12428. Epub 2018 Oct 9. PMID 30298560
- [Background] Sergl HG, Klages U, Zentner A. Pain and discomfort during orthodontic treatment: causative factors and effects on compliance. Am J Orthod Dentofacial Orthop. 1998 Dec;114(6):684-91. doi: 10.1016/s0889-5406(98)70201-x. PMID 9844209
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984
- [Background] Almallah MM, Almahdi WH, Hajeer MY. Evaluation of Low Level Laser Therapy on Pain Perception Following Orthodontic Elastomeric Separation: A Randomized Controlled Trial. J Clin Diagn Res. 2016 Nov;10(11):ZC23-ZC28. doi: 10.7860/JCDR/2016/22813.8804. Epub 2016 Nov 1. PMID 28050498
- [Background] Khattab TZ, Farah H, Al-Sabbagh R, Hajeer MY, Haj-Hamed Y. Speech performance and oral impairments with lingual and labial orthodontic appliances in the first stage of fixed treatment. Angle Orthod. 2013 May;83(3):519-26. doi: 10.2319/073112-619.1. Epub 2012 Oct 18. PMID 23075062
- [Background] Feldmann I, Bazargani F. Pain and discomfort during the first week of rapid maxillary expansion (RME) using two different RME appliances: A randomized controlled trial. Angle Orthod. 2017 May;87(3):391-396. doi: 10.2319/091216-686.1. Epub 2016 Dec 28. PMID 28029266
- [Background] Baldini A, Nota A, Santariello C, Assi V, Ballanti F, Cozza P. Influence of activation protocol on perceived pain during rapid maxillary expansion. Angle Orthod. 2015 Nov;85(6):1015-20. doi: 10.2319/112114-833.1. Epub 2015 Mar 10. PMID 25757063
- [Result] Bucci R, D'Anto V, Rongo R, Valletta R, Martina R, Michelotti A. Dental and skeletal effects of palatal expansion techniques: a systematic review of the current evidence from systematic reviews and meta-analyses. J Oral Rehabil. 2016 Jul;43(7):543-64. doi: 10.1111/joor.12393. Epub 2016 Mar 23. PMID 27004835